CLINICAL TRIAL: NCT00537953
Title: EFFICACY AND SAFETY OF A SHORT COURSE OF THE COMBINATION OF MILTEFOSINE AND ANTIMONY TO TREAT CUTANEOUS LEISHMANIASIS IN BOLIVIA
Brief Title: Short Course of Miltefosine and Antimony to Treat Cutaneous Leishmaniasis in Bolivia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Investigaciones Bioclínicas de la Fundación Fader (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-Bol/LC-1339
Record Dates: First submitted 2007-09-28; First posted 2007-10-02 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-09

CONDITIONS: Cutaneous Leihmaniasis
Keywords: Leishmaniasis; Cutaneous leishmaniasis; Miltefosine; Glucantime; Antimony; Pentavalent antimonials; Combination therapy
MeSH Terms: conditions — Leishmaniasis; Leishmaniasis, Cutaneous | interventions — miltefosine; Meglumine Antimoniate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Miltefosine , meglumine antimoniate

SUMMARY:
The combination of a half-course of miltefosine and a half-course of antimony will be evaluated for efficacy and tolerance. The combination of miltefosine and antimony is chosen because these are now the two standard agents in Bolivia, and in vitro the combination was additive to mildly synergistic against a standard leishmania strain.

DETAILED DESCRIPTION:
Combination therapy is now being used for many infectious diseases, such as tuberculosis, malaria, and HIV. Combination therapy offers the potential of preventing drug resistance, because organisms resistant to one of the drugs may be susceptible to the other drug; and also the potential to diminish drug therapy duration and thus side effects. These two potential benefits to some extent contradict each other: preventing resistance is best done if full courses of both drugs is used; diminishing therapy duration means using less than the full course of each drug. The optimum combination regimen is one in which sufficient amounts of both drugs are used to have high efficacy, yet the amounts are as low as possible to spare patients unnecessarily long courses of drug.

Until recently, the standard treatment for the leishmaniases was pentavalent antimony (Glucantime or Pentostam). The cure rate for L panamensis in Colombia is 91%-93% [Soto, 1993; Velez, 1997] and the cure rate in Bolivia, in work soon to be completed, is also 90% [ Soto, unpublished results]. A large study with several formulations of antimony found a combined Bolivia-Colombia cure rate of 86% [Soto, 2004b]. Nevertheless, pentavalent antimonials have the disadvantages of multiple injections and mild-moderate clinical toxicity [gastrointestinal complaints, liver enzyme elevations, pancreatic enzyme elevations], all of which are particularly unpleasant for a moderate clinical problem such as cutaneous leishmaniasis.

The oral agent Miltefosine has now been shown to be as effective as antimony in Colombia and Bolivia. In Colombia, the cure rate for miltefosine was 91% [Soto 2004a] and in the soon to be completed comparative trial in Bolivia, the cure rate for miltefosine appears to be 92% [Soto, unpublished results]. Side effects seen in patients with cutaneous disease that can be specifically attributed to the drug are nausea and vomiting of mild grade in approximately 25% of patients, and low-grade elevation of creatinine also in approximately 25% of patients [Soto 2001; Soto 2004]. A further disadvantage of miltefosine is that regimens shorter than 4 weeks have not been evaluated for cutaneous disease.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male Age: Adults Presentation: At least 1 lesion must be ulcerative. Parasitology: Parasitological confirmation of 1 lesion will be made by visualization or culture of leishmania from the biopsy or aspirate of the lesion.

Exclusion Criteria:

* Previous treatment for leishmaniasis, specific or putatively specific therapy (Sb, pentamidine, amphotericin B, imidazoles, allopurinol)
* Other concomitant diseases by history and by approximately normal complete blood counts (white blood count, hemoglobin, platelet count), values of liver transaminases (SGOT), values of pancreatic function (lipase), kidney function tests (creatinine), and EKG.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Berman, MD, PhD, Study Chair — AB Foundation for Medical Research; Jorge Vargas, MD, Principal Investigator — Cenetrop
Locations (1):
- Hospital Dermatológico, Jorochito, Santa Cruz Department, Bolivia